CLINICAL TRIAL: NCT02342717
Title: Relative Bioavailability of a Single Oral Dose of BI 425809 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, Two-period, Fixed-sequence Trial)
Brief Title: Relative Bioavailability of a Single Oral Dose of BI 425809 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346.10; 2014-004855-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809; Itraconazole

ARMS (2):
- Reference (Experimental): single dose BI 425809
  Interventions: Drug: BI 425809
- Test (Experimental): multiple doses of Itraconazole + single dose BI 425809
  Interventions: Drug: BI 425809; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 425809 — single dose BI 425809 tablet
  Other Names: Iclepertin
  Arms: Test
Drug: Itraconazole — multiple doses of Itraconazole capsules
  Arms: Test
Drug: BI 425809 — single dose BI 425809 tablet
  Other Names: Iclepertin
  Arms: Reference

SUMMARY:
To investigate whether and to what extent co-administration of multiple doses of itraconazole affect single dose pharmacokinetics of BI 425809 in healthy male subjects

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 halflives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two month after the trial completion. Acceptable methods of contraception comprise barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive for at least two month prior trial participation)
* Known fructose intolerance, glucose-galactose malabsorption, or saccharose-isomaltase deficiency
* History of relevant liver diseases such as disturbance of liver function, jaundice, drug induced liver injury, Dubin-Johnson syndrome, Rotor syndrome, or liver tumours
* Liver enzymes (ALT, AST, GGT) above upper limit of normal at the screening examination

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
AUC0-167 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 167 h) | 8 days postdose
Cmax (maximum measured concentration of the analyte in plasma) | 15 days postdose

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 15 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1346.10.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Desch M, Wunderlich G, Goettel M, Goetz S, Liesenfeld KH, Chan TS, Rosenbrock H, Sennewald R, Link J, Keller S, Wind S. Effects of Cytochrome P450 3A4 Induction and Inhibition on the Pharmacokinetics of BI 425809, a Novel Glycine Transporter 1 Inhibitor. Eur J Drug Metab Pharmacokinet. 2022 Jan;47(1):91-103. doi: 10.1007/s13318-021-00723-y. Epub 2021 Oct 29. PMID 34716565